CLINICAL TRIAL: NCT02892214
Title: The Reciprocal Relations Between Psychosocial Characteristics and the Progression of Vestibulodynia, and the Mental Health of the Patient
Brief Title: The Reciprocal Relations Between Psychosocial Characteristics and the Progression of Vestibulodynia
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, MD, Meir Medical Center
Other Study IDs: 0089-16-COM1
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Localized Provoked Vulvodynia
MeSH Terms: interventions — Estriol; Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hypertonic pelvic muscle dysfunction: In this subgroup, pelvic floor (PF) muscles become tight and tender. Typically, the pain is much worse at 4-8 o'clock position of the vestibule with minimal or no pain in the upper vestibule.
  Interventions: Procedure: Pelvic floor physical therapy
- Hormonally mediated PVD: The pain began while taking hormonal contraceptive or other medications that affect hormones, after removal of ovaries, breastfeeding or menopause. The entire vestibule is tender and vestibular mucosa is often dry and thin.
  Interventions: Drug: estriol cream (ovestin)
- Neuroproliferative PVD: In this condition, we speculate that women have an increased number of nociceptors in the vestibular mucosa. Pain is primary and there is tenderness of the entire vestibule.
  Interventions: Procedure: Low-level-laser therapy

INTERVENTIONS:
Procedure: Pelvic floor physical therapy
  Groups: Hypertonic pelvic muscle dysfunction
Drug: estriol cream (ovestin)
  Groups: Hormonally mediated PVD
Procedure: Low-level-laser therapy
  Groups: Neuroproliferative PVD

SUMMARY:
The proposed study will evaluate how personality characteristics, cognitive factors and the emotional and behavioral responses of patients with provoked vestibulodynia (localized provoked vulvodynia) influence the natural history of the syndrome, patients' adherence to therapeutic interventions, provoked pain levels, pelvic floor rehabilitation, emotional health and sexual functioning.

DETAILED DESCRIPTION:
Provoked vestibulodynia (PVD) is the term describing a syndrome of provoked, localized allodynia of the vestibule of the vulva, not explained by another condition, and lasting more than 3 months. PVD is not a defined disease but rather a symptom. It is thought that PVD represent a group of distinct disorders that have been classified together because they produce pain in the same anatomic location.

Studies found that different factors such as genetic, inflammation, recurrent vaginitis, allergy, trauma, emotional and neural may be involved in the development of PVD.

Treatment of PVD is generally predicated on a trial and error basis, because the pathogenesis is not defined. The result is that many forms of therapeutic interventions have been used, yet the evidence remains largely inconclusive, the response rates varies considerably, and many women do not respond to any of the treatments. It is therefore important to recognize which factors mediate the syndrome's severity, and influence the effectiveness of treatments.

The proposed study will evaluate how different patients' characteristics (personality, cognitive) and responses (emotional and behavioral) influence the natural history of the syndrome and the response to treatment. The study is based on the bio-psycho-social model and the adult attachment theory, which integrates psychosocial factors to define susceptibility to acquire pain disorders and predict response to therapy. According to this model, choosing effective coping strategy during a crisis and receiving support from a spouse are vital for recovery.

The study aim to:

1. Characterize interactions between attachment patterns, personality types, cognitive factors (catastrophization, coherence, and partner's support), emotional factors (coping strategies, emotional stress and satisfaction from intimate relationship) to pain levels, pelvic floor hypertonicity, sexual function and patient's emotional health.
2. Examine whether treatments' results are influenced by personality, relationship, cognitive, emotional and behavioral characteristics of the patient.
3. Recognize factors that influence the extent of adherence to treatment.
4. Characterize patients' profile in regard to successful outcome.

Methods Patients will be recruited from the clinic for vulvovaginal disorders in Clalit Healthcare services in Jerusalem. The diagnostic procedures, patients' sub-classification and the proposed treatments in the current protocol are identical to those currently used in the clinic. Each patient will undergo a standard evaluation which includes: detailed history intake, vulvar and vaginal examination, evaluation of vestibular tenderness (Q tip test), pelvic floor musculature tenderness examination, vaginal pH measurement, saline and 10% potassium hydroxide microscopy, yeast and bacterial cultures and STD screening.

Patients who fulfill diagnostic criteria of PVD and who will be willing to participate in the study will be asked to sign an informed consent and complete the following self-administered intake questionnaires:

* Socio-demographic questionnaire (age, marital status, religios, PVD onset, health status, education etc.)
* Close Relations Experiences questionnaire
* Five Factor Inventory -NEO-FFI
* Pain catastrophizing questionnaire
* Sense of Coherence Scale
* Ways of giving support questionnaire
* COPE -Multidimensional Coping Inventory
* Semantic Differential Measure of Marital Satisfaction
* PSS-10 - Perceived Stress Scale
* FSFI-Female Sexual Function Index

Instructions for treatment will be given in regards to the diagnosis. Patients will be instructed to schedule follow-up appointments at 3,6,9, and 12 months. During follow-up appointments they will be assessed in regard to vestibular tenderness (using various parameters), as well as by the same questionnaires. Additional treatment will be recommended according to medical status, in an identical way to this routinely used in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. A history of 3 months or more of vulvar pain suggestive of PVD, i.e. symptoms of pain on vaginal penetration (insertional dyspareunia and/or pain with tampon insertion).
2. On exam, tenderness localized within the vestibule when being touched with a cotton-tip applicator.
3. No identifiable cause for the pain, such as vulvovaginal candidiasis, vaginal atrophy, desquamative inflammatory vaginitis (DIV), herpes, dermatitis or vulvar dystrophy.

Exclusion Criteria:

1. other causes for vulvar pain
2. pregnancy or a planned pregnancy in the upcoming year
3. diagnosis of chronic disease that may affect central nervous system or general function.
4. usage of psychiatric medications or those affecting pain modulation.
5. unprovoked or mixed vulvodynia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the clinic for vulvovaginal disorders in Clalit Healthcare services in Jerusalem.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change of measure of Q tip test assessing pain intensity | Change in measure between recruitment to 3 months, 6 months , 9 months and 12 months
  The exam is performed by touching the vestibule with a cotton-tip applicator in 6 defined points (2,5,6,7, 10 and 12),while the patient is being asked to rate the intensity of pain verbally from 0 to 10 at each point.

SECONDARY OUTCOMES:
Measurement of vestibular tenderness using a vulvar algesiometer | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months.
Change of pain using Visual analog scale | Change in VAS between recruitment to 3 months, 6 months , 9 months and 12 months
Adherence to therapy | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months.
  Adherence to therapy will be assessed by calculating attendance to planed appointments (physical therapy, medical appointments and LLL treatments)
Female sexual function index questionnaire | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months.
Pelvic floor hypertonicity measurements | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months.
  Pelvic floor muscle tonicity will be evaluated using manual palpation of the muscles by the physician.
Brief Symptom Inventory-18 questionnaire (evaluating emotional symptoms) | Every 3 months for 1 year- 0, 3 months, 6 months, 9 months and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Merkaz Briot Haisha, Ramat Eshkol, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews JC. Vulvodynia interventions--systematic review and evidence grading. Obstet Gynecol Surv. 2011 May;66(5):299-315. doi: 10.1097/OGX.0b013e3182277fb7. PMID 21794194
- [Background] Antonovsky, A. (1987). How people manage stress and stay well. San Francisco, CA, US: Jossey-Bass Unraveling the mystery of health.
- [Background] Bergeron S, Binik YM, Khalife S, Pagidas K, Glazer HI, Meana M, Amsel R. A randomized comparison of group cognitive--behavioral therapy, surface electromyographic biofeedback, and vestibulectomy in the treatment of dyspareunia resulting from vulvar vestibulitis. Pain. 2001 Apr;91(3):297-306. doi: 10.1016/S0304-3959(00)00449-8. PMID 11275387
- [Background] Bergeron S, Brown C, Lord MJ, Oala M, Binik YM, Khalife S. Physical therapy for vulvar vestibulitis syndrome: a retrospective study. J Sex Marital Ther. 2002 May-Jun;28(3):183-92. doi: 10.1080/009262302760328226. PMID 11995597
- [Background] Brennan, K.A., Clark, C.L., & Shaver P.R. (1998). Self-report measurement of adult attachment: An integrative overview. In J.A. Simpson & W.S. Rholes (Eds.), Attachment theory and close relationships, (pp. 46-76). NY,US: Guilford Press.
- [Background] Buunk, B. P., Berkhuysen, M. A., Sanderman, R., Nieuwland, W., & Ranchor, A. V. (1996). Active engagement, protective buffering and overprotection: Instruments to measure the role of the spouse in heart rehabilitation. Gedrag & Gezondheid, 24, 304- 113.
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Cohen, S., & Spacapan, S. (1978). The aftereffects of stress: An attentional interpretation. Environmental Psychology and Nonverbal Behavior, 3(1), 43-57.
- [Background] Meredith P, Ownsworth T, Strong J. A review of the evidence linking adult attachment theory and chronic pain: presenting a conceptual model. Clin Psychol Rev. 2008 Mar;28(3):407-29. doi: 10.1016/j.cpr.2007.07.009. Epub 2007 Jul 19. PMID 17719157
- [Background] Sadownik LA. Clinical profile of vulvodynia patients. A prospective study of 300 patients. J Reprod Med. 2000 Aug;45(8):679-84. PMID 10986689
- [Background] Sullivan, M. J. L., Bishop, S., & Pivic, J. (1995). The pain catastrophizing scale: Development and validation. Psychological Assessment, 7, 524-532.